CLINICAL TRIAL: NCT05651100
Title: Phase 1/Phase 2 Study of Sequential Chimeric Antigen Receptor T Cell Targeting at CD19 and CD22 B-cell Antigens Treating Refractory or Relapsed B-cell Lymphoma Patients
Brief Title: Safety and Efficacy of Sequential CD19 and CD22 Targeted CAR-T Therapy for Relapsed/Refractory B Cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kecellitics Biotech Company Ltd (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kece-4
Record Dates: First submitted 2022-11-26; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Lymphoma, B-Cell
Keywords: CAR-T; Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — Antigens, CD19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm 1 (Experimental): sequential CD19 and CD22 targeted CAR-T cells treat
  Interventions: Biological: CD19 and CD22 targeted CAR-T cells

INTERVENTIONS:
Biological: CD19 and CD22 targeted CAR-T cells — CAR-T cells were manufactured from peripheral blood mononuclear cells collected by leukapheresis and frozen for multiple uses. Before each CAR T-cell infusion (day 0), patients received lymphodepleting chemotherapy composing of Fludarabine (30 mg/m2/day) and Cyclophosphamide (300 mg/m2/day) on days -5 to -3. No bridging chemotherapy was given between enrollment and infusion. In sequential CAR-T clinical trials, CAR-T cells will be given.（anti-CD19 CAR-T first, then anti-CD22 CAR-T).

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of Sequential CD19 and CD22 targeted CAR-T cells therapy for patients with relapsed/refractory B Cell Lymphoma.

DETAILED DESCRIPTION:
Although the CD19 targeted CAR-T cell therapies have gained significant results in patients with relapsed and refractory B-cell Leukemia and Lymphoma. There are some patients who resisted anti-CD19 CAR-T cells or get CD19 negative relapse. To make further improvement, We launch such a clinical trial using sequential CD19 and CD22 targeted CAR-T cells for patients with relapsed and refractory B Cell Lymphoma to evaluate the efficacy and safety of sequential CD19 and CD22 targeted CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory B cell non-hodgkin lymphoma.
2. KPS>60.
3. Life expectancy>12 weeks.
4. Gender unlimited, age from 3 years to 70 years.
5. Evidence for cell membrane CD19 and/or CD22 expression;
6. Patients who have failed at least one line of a standard treatment.
7. No serious mental disorder.
8. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
9. No other serious diseases(autoimmune disease, immunodeficiency etc.).
10. No other tumors.
11. Patients volunteer to participate in the research.
12. Patients with history of allogeneic stem cell transplantation are eligible if at least 100 days post-transplant, if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to trial

Exclusion Criteria:

1. Pregnancy and nursing females.
2. Patients are allergic to cytokines.
3. Uncontrolled active infection.
4. Acute or chronic GVHD.
5. Treated with T cell inhibitor.
6. Patients who had used steroid hormones within one week.
7. Patients who had used Rituximab within two weeks.
8. HIV/HBV/HCV Infection.
9. Other situations we think improper for the research.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 1 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Overall remission rate (ORR) | 3 months
  The ORR of Sequential CD19 and CD22 CAR-T treatment will be recorded and assessed according to the revised 2014 Lugano Criteria.

SECONDARY OUTCOMES:
complete response(CR) | 24 months
  The CR of Sequential CD19 and CD22 CAR-T treatment will be recorded and assessed according to the revised 2014 Lugano Criteria.
partial response(PR) | 24 months
  The PR of Sequential CD19 and CD22 CAR-T treatment will be recorded and assessed according to the revised 2014 Lugano Criteria.
stable disease(SD) | 24 months
  The SD of Sequential CD19 and CD22 CAR-T treatment will be recorded and assessed according to the revised 2014 Lugano Criteria.
progressive disease(PD) | 24 months
  The PD of Sequential CD19 and CD22 CAR-T treatment will be recorded and assessed according to the revised 2014 Lugano Criteria.
Duration of remission (DOR) | 24 months
  DOR will be assessed from the first assessment of CR/CRi to the first assessment of recurrence or progression of the disease or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: li xiangqun, doctor, Study Chair — Kecellitics Biotech Company Ltd
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China